CLINICAL TRIAL: NCT06587139
Title: An Online Mentoring Program to Prevent Adversities Among Trans and Other Gender Minority Youth (PILOT RCT PHASE)
Brief Title: Evaluation of Teen Connection Project for Trans and Gender Minority Youth
Acronym: TCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Rhode Island (Other)
Responsible Party: Principal Investigator, Katie M Edwards, Professor, School of Social Work Director, Interpersonal Violence Research Laboratory (IVRL), University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23676
Record Dates: First submitted 2024-08-09; First posted 2024-09-19 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Recreational Drug Use; Sexual Violence; Victimisation; Depressive Symptoms; Anxiety; Suicidal Ideation; Risk-Taking; Alcohol Drinking
Keywords: Risk-Taking; Sexual Behavior; Sex Offenses; Intimate Partner Violence; Crime Victims
MeSH Terms: conditions — Recreational Drug Use; Depression; Anxiety Disorders; Suicidal Ideation; Risk-Taking; Alcohol Drinking; Sexual Behavior

STUDY DESIGN:
Intervention Model Description: transgender and/or gender minority youth (TGMY) (n=80) are randomly assigned to a treatment (n=40) or wait-list (n=40) control condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment (Experimental): The Teen Connection Project (TCP) is theoretically grounded, and follows best practices for effective health behavior prevention. It includes seven 90-minute sessions with group and one-on-one mentoring components. The intervention is facilitated by transgender and/or gender minority adults (i.e., any identity other than cisgender).
  Interventions: Behavioral: Teen Connection Project (TCP)
- Waitlist control (No Intervention): Provide check-ins, provide resources, and offer program after intervention and measurement has been completed.
- Mentors (No Intervention): Mentors complete a two-day training and post-training survey, facilitate programming, and complete post-session surveys. A subset of the mentors will complete exit interviews.

INTERVENTIONS:
Behavioral: Teen Connection Project (TCP) — The Teen Connection Project (TCP) includes seven 90-minute sessions facilitated by transgender and/or gender minority (TGM) adults. Each transgender and/or gender minority youth (TGMY) will be paired with a TGM adult mentor based on TGMYs' rank-ordered preference for mentors. The research team seeks to match mentors & mentees such that each TGMY is matched with one of their top 3 preferred mentors. Mentors and mentees participate together in each session along with other mentors & mentees. Facilitators direct activities/discussion to promote TGMY social-emotional skills acquisition and facilitate mentor-mentee conversations. TCP sessions also include mentor-mentee breakout sessions where mentors share challenges they personally faced as TGMY and how they overcame them. Break-out discussions focus on self-acceptance, coming out, dating questions, hopes and goals for the future, & how other marginalized social identities, such as race and ethnicity, intersect with identifying as TGMY.
  Other Names: TCP
  Arms: Treatment

SUMMARY:
The purpose of this project is to develop and evaluate an online mentoring and skill-building program for transgender and/or gender minority youth (TGMY) ages 14 to 18, the Teen Connection Project (TCP). The TCP includes seven 90-minute sessions facilitated by transgender and/or gender minority (TGM) adults (who are also mentors). TGMY will be paired with a TGM adult mentor, based on their shared interests. Mentors and mentees will participate together in each session along with other mentors and mentees. Mentors will direct activities and discussion to promote TGMY social-emotional skills. The TCP sessions will include one-on-one mentor-mentee break-out sessions.

DETAILED DESCRIPTION:
Transgender and/or gender minority youth (TGMY) (i.e., any identity other than cisgender) experience concerning rates of mental health problems, self-harm, alcohol and drug use, sexual risk-taking, and violence victimization and perpetration. Minority stress theory states that peer and family rejection and internalized transphobia predict negative health outcomes in TGMY. This highlights the urgent need to identify effective programs that prevent psychosocial and behavioral health issues among TGMY. Mentoring programs may be especially impactful for TGMY, given that these programs may help alleviate adverse outcomes associated with peer and family rejection, and promote self-acceptance among TGMY. However, few mentoring programs exist specifically for TGMY, and those that do have not been rigorously evaluated; often require guardian permission; generally occur in person via community organizations--which excludes TGMY in high stigma, rural areas of the United States from participating; and rarely include evidence-based skill-building components (e.g., social-emotional skills).

The specific aims of this trial are as follow:

1. Assess acceptability and feasibility of the Teen Connection Project (TCP) through observations (to evaluate program delivery and observe mentor-mentee interactions), post-session surveys, and exit interviews with participants.
2. Generate preliminary data on the TCP's efficacy in reducing psychosocial and behavioral health issues facing TGMY, including mental health problems, self-harm, alcohol and drug use, sexual risk-taking, and teen dating violence.
3. Identify treatment options for TGMY.

The purpose of this project is to develop and evaluate an online mentoring and skill-building program for transgender and/or gender minority youth (TGMY) ages 14 to 18, the Teen Connection Project (TCP). The TCP includes seven 90-minute sessions facilitated by transgender and/or gender minority (TGM) adults (who are also mentors). TGMY will be paired with a TGM adult mentors, based on their shared interests. Mentors and mentees will participate together in each session, along with other mentors and mentees. Mentors will direct activities and discussion to promote TGMY social-emotional skills. The TCP sessions will include one-on-one mentor-mentee break-out sessions.

ELIGIBILITY:
Inclusion Criteria for Youth:

* identify as transgender and/or gender minority youth (TGMY) (i.e., any identity other than cisgender)
* be between the ages of 14 to 18 years
* read and speak English
* live in the United States
* report consistent access to a phone, tablet, and/or computer with high-speed internet access/Wi-Fi (which represents 90+% of youth in the United States)
* report an ability to attend seven, 90-minute online sessions at pre-determined times
* pass an assent quiz
* report moderate to high levels of internalized transphobia

Exclusion Criteria for Youth:

* be at imminent risk for suicide (e.g., intent to kill themselves in the immediate future) as determined by an initial online suicide screening regarding their past month suicide risk (the Suicide Behaviors Questionnaire-Revised [SBQ-R]; modified to assess past month risk)
* demonstrate current psychosis as determined by the Prodromal Questionnaire; modified to just focus on visual and auditory symptoms

Inclusion Criteria for Mentors:

* be 30 years old or older
* identify as transgender and/or gender minority (i.e., any identity other than cisgender)

Exclusion Criteria for Mentors:

• not be currently experiencing substance use disorder or mental health challenges

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Transgender and/or gender minority (i.e., any identity other than cisgender)
Enrollment: 56 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Alcohol Use (Youth-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention), Time 3 (3 months post-intervention)
  Youth Risk Behavior Survey Questionnaire (YRBSS). Minimum Value = 0, Maximum Value = 6, Higher scores = worse outcomes
Drug Use (Youth-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention), Time 3 (3 months post-intervention)
  YRBSS. Minimum Value = 0, Maximum Value = 5, Higher scores = worse outcomes
Sexual Risk-Taking (Youth-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention), Time 3 (3 months post-intervention)
  Researcher-created items, adapted items with input from a youth advisory board from, YRBSS, and Sexual Risk Taking Survey. Minimum Value = 1, Maximum Value = 7, Higher scores = worse outcomes
Dating and Sexual Violence (DSV) victimization-1 (Youth-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention), Time 3 (3 months post-intervention)
  Measure of Adolescent Relationship Harassment and Abuse (MARSHA). Minimum Value = 0, Maximum Value = 3, Higher scores = worse outcomes
DSV perpetration-1 (Youth-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention), Time 3 (3 months post-intervention)
  MARSHA. Minimum Value = 0, Maximum Value = 3, Higher scores = worse outcomes
DSV victimization-2 (Youth-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention), Time 3 (3 months post-intervention)
  CTS-2: SGM-Specific Intimate partner Violence (IPV) Tactics Scale [CTS = Conflict Tactics Scale, SGM = sexual and gender minority]. Minimum Value = 0, Maximum value = 3, Higher scores = worse outcomes
DSV perpetration-2 (Youth-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention), Time 3 (3 months post-intervention)
  CTS-2: SGM-Specific IPV Tactics Scale. Minimum Value = 0, Maximum Value = 3, Higher scores = Worse outcomes
Depressive symptoms (Youth-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention), Time 3 (3 months post-intervention)
  Patient Health Questionnaire for Adolescents (PHQ-9). Minimum Value = 0, Maximum Value = 3, Higher scores = Worse outcomes
Anxiety symptoms (Youth-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention), Time 3 (3 months post-intervention)
  Generalized Anxiety Disorder Screener (GAD-7). Minimum Value = 0, Maximum Value = 3, Higher scores = Worse outcomes
Suicidality (Youth-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention), Time 3 (3 months post-intervention)
  Suicidal Ideation Attributes Scale (SIDAS). Minimum Value = 0, Maximum Value = 10, Higher scores = Better outcomes

OTHER OUTCOMES:
Social-Emotional Competence (Youth-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention), Time 3 (3 months post-intervention)
  Social-Emotional Competence Questionnaire (SEC-Q). Minimum Value = 1, Maximum Value = 6, Higher scores = Better outcomes
Gender Minority Stress (Youth-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention), Time 3 (3 months post-intervention)
  Gender Minority Stress and Resilience Scale (adolescent extension version). Minimum Value = 1, Maximum Value = 5, Higher scores = Worse outcomes
Outness (Youth-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention), Time 3 (3 months post-intervention)
  Nebraska Outness Scale, Minimum Value = 0, Maximum Value = 100, Higher scores = Better outcomes
Positive Identity (Youth-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention), Time 3 (3 months post-intervention)
  Lesbian, Gay, and Bisexual Positive Identity Measure. Minimum Value = 1, Maximum Value = 7, Higher scores = Better outcomes
Hope for the Future (Youth-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention), Time 3 (3 months post-intervention)
  Feelings about being LGBTQIA2+. Minimum Value = 1, Maximum Value = 4, Higher scores = Better outcomes
Mentor Process Scale (Adult-reported) | Time 1 (baseline, pre-intervention), Time 2 (immediately post-intervention)
  The Mentor Process Scale consists of three subscales (Role Modeling and Identification, Relationship and Emotional Support, Teaching and Information Providing) from which survey items are drawn and minimally adapted. Minimum Value = 1, Maximum Value = 7, Higher scores = Better outcomes
Reflection and Evaluation (Adult-reported) | Time 2 (immediately post-intervention)
  Mentors' reflections and feedback are collected using an adaptation of Keller et al. (2022)'s implementation evaluation scale. Minimum Value = 1, Maximum Value = 5, Higher scores = Better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Katie M Edwards, PhD, Principal Investigator — University of Michigan
Locations (1):
- [online program, administered by the University of Nebraska-Lincoln], Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
This data will not be shared publicly. However, the PI intends to share the aggregated, de-identified quantitative survey data if users commit to the following: (a) using the data only for research purposes and not to identify any individual participant; (b) securing the data using appropriate computer technology; and (c) destroying or returning the data after analyses are completed. If the researcher agrees, in writing, to these stipulations, the PI will send them (via a link to a secure UNL OneDrive folder) the dataset prepared using SPSS (latest version available).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available in December of 2025. It will be available for 7 years until December of 2032.
Access Criteria: The PI intends to share the aggregated, de-identified quantitative survey data if users commit to the following: (a) using the data only for research purposes and not to identify any individual participant; (b) securing the data using appropriate computer technology; and (c) destroying or returning the data after analyses are completed. If the researcher agrees, in writing, to these stipulations, the PI will send him/her the dataset prepared using SPSS 24.0 (or the latest version available). The prepared data set will not include identifying information from any participant. The master list will be destroyed as soon as participants' data are linked across time. Research participants will be identified by number. A detailed codebook will be prepared and supplied with the data indicating information about each variable as well as how composite scale scores are calculated. The syntax for any data imputations will also be provided.

REFERENCES:
- [Background] CDC (2023). Youth Risk Behavior Survey. Centers for Disease Control and Prevention. https://www.cdc.gov/healthyyouth/data/yrbs/index.htm
- [Background] Turchik JA, Garske JP. Measurement of sexual risk taking among college students. Arch Sex Behav. 2009 Dec;38(6):936-48. doi: 10.1007/s10508-008-9388-z. Epub 2008 Jun 19. PMID 18563548
- [Background] Rothman EF, Cuevas CA, Mumford EA, Bahrami E, Taylor BG. The Psychometric Properties of the Measure of Adolescent Relationship Harassment and Abuse (MARSHA) With a Nationally Representative Sample of U.S. Youth. J Interpers Violence. 2022 Jun;37(11-12):NP9712-NP9737. doi: 10.1177/0886260520985480. Epub 2021 Jan 5. PMID 33399026
- [Background] Rothman EF, Paruk J, Cuevas CA, Temple JR, Gonzales K. The Development of the Measure of Adolescent Relationship Harassment and Abuse (MARSHA): Input From Black and Multiracial, Latinx, Native American, and LGBTQ+ Youth. J Interpers Violence. 2022 Mar;37(5-6):2126-2149. doi: 10.1177/0886260520936367. Epub 2020 Jul 5. PMID 32627640
- [Background] Dyar C, Messinger AM, Newcomb ME, Byck GR, Dunlap P, Whitton SW. Development and Initial Validation of Three Culturally Sensitive Measures of Intimate Partner Violence for Sexual and Gender Minority Populations. J Interpers Violence. 2021 Aug;36(15-16):NP8824-NP8851. doi: 10.1177/0886260519846856. Epub 2019 May 5. PMID 31057032
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Richardson LP, McCauley E, Grossman DC, McCarty CA, Richards J, Russo JE, Rockhill C, Katon W. Evaluation of the Patient Health Questionnaire-9 Item for detecting major depression among adolescents. Pediatrics. 2010 Dec;126(6):1117-23. doi: 10.1542/peds.2010-0852. Epub 2010 Nov 1. PMID 21041282
- [Background] van Spijker BA, Batterham PJ, Calear AL, Farrer L, Christensen H, Reynolds J, Kerkhof AJ. The suicidal ideation attributes scale (SIDAS): Community-based validation study of a new scale for the measurement of suicidal ideation. Suicide Life Threat Behav. 2014 Aug;44(4):408-19. doi: 10.1111/sltb.12084. Epub 2014 Feb 24. PMID 24612048
- [Background] Zhou M, Ee J. Development and validation of the Social Emotional Competence Questionnaire (SECQ). The International Journal of Emotional Education. 2012;4(2):27-42.
- [Background] Hidalgo MA, Petras H, Chen D, Chodzen G. The Gender Minority Stress and Resilience Measure: Psychometric Validity of an Adolescent Extension. Clin Pract Pediatr Psychol. 2019;7(3):278-290. doi: 10.1037/cpp0000297. PMID 33224698
- [Background] Meidlinger, P. C., & Hope, D. A. (2014). Differentiating disclosure and concealment in measurement of outness for sexual minorities: The Nebraska Outness Scale. Psychology of Sexual Orientation and Gender Diversity, 1(4), 489.
- [Background] Riggle, E. D., Mohr, J. J., Rostosky, S. S., Fingerhut, A. W., & Balsam, K. F. (2014). A multifactor lesbian, gay, and bisexual positive identity measure (LGB-PIM). Psychology of Sexual Orientation and Gender Diversity, 1(4), 398.
- [Background] University of Connecticut and the Human Rights Campaign. 2022 National Survey on LGBTQ Youth Mental Health. https://www.thetrevorproject.org/survey-2022/
- [Background] Turchik JA, Garske JP. Sexual risk survey. In: Fisher TD, Davis CM, Yarber WL, Davis SL, eds. Handbook of sexuality-related measures. 3rd ed. Routledge; 2010:600-602.
- [Background] Tolan PH, McDaniel HL, Richardson M, Arkin N, Augenstern J, DuBois DL. Improving understanding of how mentoring works: Measuring multiple intervention processes. J Community Psychol. 2020 Aug;48(6):2086-2107. doi: 10.1002/jcop.22408. Epub 2020 Jul 11. PMID 32652575
- [Background] Keller TE, Drew AL, Herrera C, Clark-Shim H, Spencer R. Do program practices matter for mentors?: How implementation of empirically supported program practices is associated with youth mentoring relationship quality. J Community Psychol. 2023 Nov;51(8):3194-3215. doi: 10.1002/jcop.23019. Epub 2023 Feb 25. PMID 36840743

DOCUMENTS (1):
  • Informed Consent Form (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT06587139/ICF_000.pdf